CLINICAL TRIAL: NCT05946889
Title: Comparisons of Human Fibrin Glue (Tisseel) Versus Suture and Robotic Versus Traditional Laparoscopy for Ovarian Cystectomy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 111192-E
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: Women With Ovarian Cyst

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suture: Women with ovarian cyst who received robotic/laparoscopic ovarian cystectomy with suture
- Human Fibrin Glue: Women with ovarian cyst who received robotic/laparoscopic ovarian cystectomy with human fibrin glue

SUMMARY:
Objective: To compare the effects of suture versus human fibrin glue during robotic or laparoscopic ovarian cystectomy

DETAILED DESCRIPTION:
Methods: The medical records of all consecutive women who received robotic or laparoscopic ovarian cystectomy between January 2016 and May 2022 were reviewed. Perioperative outcome and ovarian size were compared.

Expected results: We can get the effects of suture versus human fibrin glue during robotic or laparoscopic ovarian cystectomy. The above information should be important for consultation.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old women
* women who received robotic or laparoscopic ovarian cystectomy between January 2016 and May 2022 were reviewed.

Exclusion Criteria:

* Patients who underwent myomectomy at the same time.

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — ovarian cystectomy
Study Population: Patients who received ovarian cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Ovarian size | 24 months
  the ovarian size after ovarian cystectomy during follow-up

SECONDARY OUTCOMES:
Blood loss | 1 week
  Estimated blood loss during perioperative period (including abdominal drainage)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan